CLINICAL TRIAL: NCT00005400
Title: Angiotensinogen Variants and Adverse Pregnancy Outcomes
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4317; R01HL055812 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-01-21 (Estimated); Status verified 2016-01

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Pre-Eclampsia
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Pre-Eclampsia

SUMMARY:
To examine angiotensinogen genetic variants and adverse pregnancy outcomes.

DETAILED DESCRIPTION:
BACKGROUND:

Early in gestation maternal blood volume normally expands by an unknown mechanism; failure of this normal adaptation to pregnancy has been associated with common adverse pregnancy outcomes including preeclampsia, intrauterine growth retardation, and premature labor. The renin-angiotensin system has a critical role in controlling maternal fluid volume and probably in the pathophysiology of these serious complications of pregnancy. Kenneth Ward and his group have recently discovered DNA variants which cause amino acid substitutions in angiotensinogen (renin substrate), one of which (T235) is strongly associated with preeclampsia. They hypothesize that functionally different angiotensinogen proteins may underlie the pathophysiology of preeclampsia and other related disorders (such as intrauterine growth retardation and premature labor) by not allowing normal volume expansion to occur.

The four interrelated approaches in the study should lead to a better understanding of the role of angiotensinogen in pregnancy and of the pathophysiology of preeclampsia. Unlike any previous finding in preeclamptic patients, the genetic alteration in angiotensinogen described is an intrinsic defect which, although it may be modified by other factors, cannot be 'secondary' to other pathophysiologic variables. This molecular hypothesis demands a reinterpretation of many prior findings in preeclampsia, fetal growth retardation, and premature labor based on angiotensinogen genotypes. The DNA and plasma collected for this study will be invaluable resources for future molecular investigations of abnormal pregnancies.

DESIGN NARRATIVE:

Four different strategies were used. First, a prospective, epidemiologic survey of 24,000 pregnancies was conducted to determine the role of the T235 variant in common disorders of pregnancy. From this population, nulligravida volunteers, 150 who were homozygous for T235 variant and 150 who were homozygous for the alternative M235 allele, were selected for a longitudinal study of maternal-fetal physiology and biochemistry in order to determine how and when the T235 variant exerted its adverse effect. Taking advantage of the large average family size in Utah, the female relatives of women with preeclampsia were also studied in order to define the genetics of important angiotensinogen variants. Finally, DNA from preeclamptic patients was examined for additional mutations in the angiotensinogen gene which may offer unique pathophysiologic insight.

The study was renewed in 1999 for another four years to investigate the hypothesis that disease-associated angiotensinogen alleles promote abnormal spiral artery remodeling and inhibit maternal plasma volume expansion.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1995-08; Study Completion 2003-07

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Ward — University of Utah